CLINICAL TRIAL: NCT01572818
Title: Effects of Phlebotomy on Insulin Sensitivity in Insulin Resistance-associated Hepatic Iron Overload Patients
Acronym: SAINPOS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rennes University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008-A00636-49; PHRC/07-05 (Other: Rennes University Hospital); CIC0203/070 (Other: Center for Clinical Research of Rennes)
Record Dates: First submitted 2011-05-17; First posted 2012-04-06 (Estimated); Last update posted 2016-06-15 (Estimated); Status verified 2016-06

CONDITIONS: Insulin Resistance; Iron Overload
Keywords: Phlebotomy; Insulin Resistance; Iron Overload
MeSH Terms: conditions — Insulin Resistance; Iron Overload | interventions — Phlebotomy; Diet

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Phlebotomy (Experimental): phlebotomy associated with dietary and lifestyle counseling
  Interventions: Procedure: phlebotomy; Behavioral: dietary and lifestyle counseling
- Lifestyle counseling (Active Comparator): dietary and lifestyle counseling
  Interventions: Behavioral: dietary and lifestyle counseling

INTERVENTIONS:
Procedure: phlebotomy — 7 ml/kg without exceeding 500 mL
  Other Names: Non applicable.
  Arms: Phlebotomy
Behavioral: dietary and lifestyle counseling — dietary and lifestyle counseling
  Other Names: Non applicable.

SUMMARY:
The purpose of this study is to evaluate efficacy of phlebotomy on insulin sensitivity as evaluated by euglycemic-hyperinsulinic clamp in insulin resistance-associated hepatic iron overload patients.

DETAILED DESCRIPTION:
The main objective of this study is to evaluate in patients with HSD effects of treatment with phlebotomy rules with lifestyle and dietary rules versus lifestyle modifications alone on peripheral insulin resistance (assessed by hyperinsulinemic clamp).

Secondary objectives are:

* to study in all patients with HSD the relationship between the amount of iron intrahepatic and degree of peripheral insulin resistance and liver before therapeutic intervention.
* to study and compare the effects of phlebotomy treatment versus no treatment on:

  * Plasma levels of adipocytokines,
  * Plasma concentrations of inflammatory markers and markers of insulin resistance,
  * The serum ferritin,
  * The post-hepatic clearance of insulin,
  * The surface of the abdominal visceral fat and subcutaneous abdominal.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 70 years
* Ferritin between 450 and 1000 µg/L
* Hepatic iron overload proved by MRI (CHF >36 µmol/g)
* Body mass index > 25 kg/m²
* Fasting glycemia <1,26 g/L
* HbA1c < 6,5%
* Signed written and informed consent

Exclusion Criteria:

* Other causes of hyperferritinemia:

  * Inflammatory syndrome (CRP >10 mg/L) or inflammatory, immune or malignant diseases
  * Hyperferritinemia-cataract syndrome (familial cataract or personal history of cataract before 50 years old)
  * Low ceruloplasmin level
  * Porphyria (cutaneous signs)
  * Haemochromatosis established by the genotype (C282Y homozygous or C282Y/H63D coumpound heterozygous genotypes)
* Contraindication of phlebotomy

  * Haemoglobin <13,5 g/dL (threshold established by the Etablissement Français du Sang)
  * Heart failure or coronary heart diseases
  * Hepatic failure, renal (GFR <50mL/min) or respiratory insufficiency (chronic dyspnea)
  * Poor venous system
* Viral, immune, genetic, vascular, malignant or toxic chronic hepatic disease
* Alcohol consumption more than 21 doses per week during 5 years or more
* Type 1 or type 2 diabetes
* Oral anti-diabetic, corticoids or immune suppressor drugs
* Hepatic severe disease
* Claustrophobia, having a pace-maker or intracerebral clips
* Subjects deprived of their liberty by judicial or administrative decision, subjects that are not affiliated to social security or topics exclusion period of a previous study

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2010-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Glucose Infusion Rate by euglycemic-hyperinsulinic clamp | 6 months

SECONDARY OUTCOMES:
hepatic parameters | 6 months
inflammation markers | 6 months
  IL-6, TNF alpha, CRP
Adipokins markers | 6 months
  adiponectin, PAI1, leptin
SHBG | 6 months
HOMA-IR | 6 months
Hepatic iron overload (MRI) | 6 months
  transaminase (ALT, AST), gamma GT
Abdominal and sub-cutaneous fat surface (MRI) | 6 months
iron parameters | at 6 months
  serum iron, ferritin, saturation of transferrin
lipid profile | at 6 months
  HDL-c, LDL-c, triglycerides

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice BONNET, MD, PHD, Principal Investigator — Rennes University Hospital; Eric Bellissant, MD, PhD, Study Chair — RennesUniversity Hospital
Locations (2):
- France (2):
  - CHU, Nantes
  - CHU, Rennes